CLINICAL TRIAL: NCT03194503
Title: Improving Safety and Quality of Tracheal Intubations in Neonatal ICUs
Brief Title: Tracheal Intubation Coaching in NICUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Washington (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-013606; 1R21HD089151-01A1 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-06-21 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Failed or Difficult Intubation, Sequela; Intubation;Difficult; Intubation Complication
Keywords: Intubation; Video Laryngoscope; Coaching/training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Attendings (Active Comparator): Study intervention is a VL coaching training for site neonatology attendings. Each site leader/key educator will be trained remotely by expert co-investigators. Site leaders and key educators will train their attendings. The quality of VL coaching skills will be verified by randomly auditing 20% of attending providers at each site for their skill assessment by remote simulation during the transition/post-intervention phase.
  Interventions: Device: VL Coaching training using C-MAC video laryngoscope
- Trainees (No Intervention): Trainees will be coached as usual by attendings during their supervised intubation events

INTERVENTIONS:
Device: VL Coaching training using C-MAC video laryngoscope — Each neonatology attending providers will receive a video laryngoscopy coaching training using a C-MAC video laryngoscope and an intubation training manikin available at each site by a site leader. During the training, site leader will act as a trainee confederate, and each neonatology attending provider will be trained to coach a trainee utilizing video images from C-MAC video laryngoscope and a cognitive aid with standardized language in a laminated card. This training part typically takes approximately 15-30 minutes including consenting process.
  Each site leader will be trained by PI or PI's designee using remote simulation. In this remote simulation, each site leader will coach an actor at the Children's Hospital of Philadelphia (CHOP) using a profile video image and C-MAC video laryngoscopy image through CHOP approved video conferencing software. A standardized language will be taught to each site leader with a cognitive aid (laminated card).
  Arms: Attendings

SUMMARY:
The purpose of the study is to determine the efficacy of video coaching training for neonatology attending providers on tracheal intubation procedural outcomes in neonatal ICUs.

DETAILED DESCRIPTION:
Tracheal intubation (TI) is the most common life-saving intervention for resuscitation and stabilization of critically ill neonates in Neonatal Intensive Care Units (NICUs).Recently, video laryngoscopy (VL) has become available in neonatal clinical practice to allows trainees and frontline providers to perform standard direct airway visualization (i.e., traditional laryngoscopy) while the supervisor can simultaneously view a real-time video displaying what the laryngoscopist is seeing. However, VL associated coaching during TI has not been rigorously evaluated.The purpose of the study is to determine the efficacy of video coaching training for neonatology attending providers on tracheal intubation procedural outcomes in neonatal ICUs. The primary objective of this study is to determine whether the video coaching skill training for neonatology attendings reduces the occurrence of adverse tracheal intubation associated events among all tracheal intubations in neonatal ICUs over 2 years before and after intervention. The secondary objectives are to 1) determine if video coaching training is feasible to all neonatology attending physicians using train the trainer approach with a remote simulation and 2) determine if the video coaching skill competency among neonatology attending physicians who completed the training using a remote simulation

ELIGIBILITY:
Inclusion Criteria:

1. VL coach: Neonatology attending physician position at each neonatal ICU, or Senior trainees who are anticipated to graduate within next 6 months to become neonatology attending physicians.
2. VL coach receivers: Trainees (medical students, residents, fellows except those graduating within next 6 months) and frontline providers (nurse practitioners, hospitalists, physician assistants, respiratory therapists, others who perform tracheal intubations under attending physicians' supervision)

Exclusion Criteria:

None

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akira Nishisaki, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (10):
- United States (8):
  - University of California San Diego Jacobs Medical Center, La Jolla, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - WakeMed, Raleigh, North Carolina
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- CHU Sainte-Justine, Montreal, Quebec, Canada
- KK Women's and Children's Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Intervention: Intubations before VL coaching using train-the-trainer mechanism was implemented.
- Post- Intervention: Intubations after VL coaching using train-the-trainer mechanism was implemented.
Period: Overall Study
Arm/Group | Pre-Intervention | Post- Intervention
Started | 458 | 1054
Completed | 458 | 1054
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Post-Intervention: Intubations after VL coaching using train-the-trainer mechanism was implemented.
- Total: Total of all reporting groups
Arm/Group | Pre-Intervention | Post-Intervention | Total
Number analyzed (Participants) | 458 | 1054 | 1512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 458 | 1054 | 1512
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 452 | 648
  Male | 262 | 602 | 864
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 14 | 20
  Asian | 24 | 53 | 77
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 70 | 161 | 231
  White | 329 | 759 | 1088
  More than one race | 27 | 63 | 90
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tracheal Intubation Associated Events (TIAEs) in the NICU Over 2 Years
Description: Reduction in the occurrence of adverse tracheal intubation associated events among all tracheal intubations in neonatal ICUs over 2 years after neonatology attendings receive video coaching skill training.
Time Frame: 2 years
Population: The primary outcome is comparing the number of participants with intubations before the intervention implementation phase (n=458) and the number of participants with intubations in the post intervention implementation phase (n=1,054), total n=1,512 for outcome 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 458 | 1054
Participants
  Any TIAEs | 138 | 214
  Severe TIAEs | 33 | 51
  Severe Desaturation (>20%) | 244 | 491
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; This statistical analysis applies to all three rows in the post-intervention column. ITT analysis: Multivariable analysis for Any TIAEs, Severe TIAEs, and Severe desaturation(>20%); Test type: Superiority; p = 0.015, t-test, 2 sided; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.47 to 0.92]

2. Secondary Outcome: Number of Participants With Severe Oxygen Desaturation (>20% Decline in SpO2) Among Those With VL Coaching and Without VL Coaching
Description: Intubations with VL coaching vs. no VL coaching (incl: DL&VL) can reduce severe oxygen desaturation:
  Oxygen desaturation defined as highest -lowest SpO2 during the intubation is >20% (absolute value). Intervention timing was randomized based on the site size.
Time Frame: 18 months
Population: The number of participants in this outcome measure include those intubated with VL coaching (n=155) and those intubated without VL coaching (n=984), total n=1,139 for outcome measure 2.
Measure: Count of Participants; unit: Participants
Groups:
- VL Coaching: Intubations where the intubator (trainee) was coached by an attending to use Video Laryngoscopy.
- No VL Coaching (Including DL&VL): Intubations where the intubator was not coached to use Video Laryngoscopy or direct laryngoscopy was used.
Arm/Group | VL Coaching | No VL Coaching (Including DL&VL)
Number analyzed (Participants) | 155 | 984
Participants
  Any TIAEs | 23 | 209
  Severe TIAEs | 5 | 49
  Severe Desaturation (>20%) | 99 | 438
Statistical Analysis 1: Comparison: VL Coaching vs No VL Coaching (Including DL&VL); This statistical analysis applies to all three rows and is a per-protocol analysis: Multivariable analysis for Any TIAEs, Severe TIAEs, and Severe desaturation(>20%); Test type: Superiority; p = 0.250, t-test, 2 sided; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.50 to 1.20]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 18 months from January 1, 2018 to June 30, 2019.
Description: Study procedures are not greater than minimal risk, SAE are not expected. If unanticipated problems related to the research involving risks to subjects or others happened during the course of the study (including SAEs) they would be reported to the IRB. in accordance with CHOP IRB SOP 408: Unanticipated Problems Involving Risks to Subjects. AEs that are not serious but that are notable and could involve risks to subjects will be summarized in narrative or other format and submitted to the IRB.
Arm/Group | Pre-Intervention | Post-Intervention
All-Cause Mortality (participants affected / at risk) | 0/458 | 0/1054
Serious Adverse Events (participants affected / at risk) | 0/458 | 0/1054
Other Adverse Events (participants affected / at risk) | 0/458 | 0/1054

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03194503/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03194503/ICF_001.pdf